CLINICAL TRIAL: NCT01000441
Title: Rotation or Change of Biotherapy After First Anti-TNF Treatment Failure for Rheumatoid Arthritis
Acronym: ROC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4507
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis with inadequate response to 1 anti-TNF
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab; Etanercept; Adalimumab; Abatacept; Rituximab; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- arm 1 (2d anti-TNF): (Active Comparator): infliximab, etanercept, adalimumab
  Interventions: Drug: infliximab, etanercept, adalimumab
- arm 2 (other biotherapy) (Active Comparator): abatacept, rituximab or tocilizumab
  Interventions: Drug: abatacept, rituximab or tocilizumab

INTERVENTIONS:
Drug: infliximab, etanercept, adalimumab
  Arms: arm 1 (2d anti-TNF):
Drug: abatacept, rituximab or tocilizumab
  Arms: arm 2 (other biotherapy)

SUMMARY:
Approximately 30% of patients with rheumatoid arthritis have an inadequate response to anti-TNF (primarily or loss of response), leaving two alternatives: rotation to a second anti-TNF or change of biologic, with a different mechanism of action, such as abatacept, rituximab and tocilizumab. No controlled trial compared these two strategies face to face. The present objective is to investigate the issue whether one of these strategies could have a better efficacy in a pragmatic trial in the setting of current practice.

ELIGIBILITY:
Inclusion Criteria:

* Active and erosive rheumatoid arthritis with a DAS28 equal or greater than 3.2
* Inadequate response to a 1st anti-TNF
* Stable or no treatment with any DMARDs, or oral corticosteroids (< or = to 10 mg/day of prednisone equivalent)during the preceding month

Exclusion Criteria:

* Counter-indication to other anti-TNF, abatacept, rituximab or tocilizumab
* Pregnancy
* Age < 18 years
* Impossibility to give informed consent
* Impossibility to be followed for 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-12-23 (Actual); Primary Completion 2013-08-12 (Actual); Study Completion 2013-08-12 (Actual)

PRIMARY OUTCOMES:
Proportion of EULAR responders | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacques-Eric GOTTENBERG, MD, PhD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (44):
- France (43):
  - Polyclinique de Picardie, Amiens
  - Centre Hospitalier de Belfort-Montbéliard, Belfort
  - CHU de Besançon - Hôpital Jean Minjoz, Besançon
  - Hôpital Jean Verdier, Bondy
  - CHU Bordeaux - Hôpital Pellegrin, Bordeaux
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - CHU de la Cavale Blanche, Brest
  - CHU de Caen, Caen
  - Centre Hospitalier Jean Rougié, Cahors
  - Centre Hospitalier de Cannes, Cannes
  - CHU Gabriel Montpied, Clermont-Ferrand
  - Hôpitaux Civils de Colmar, Colmar
  - CHU de Grenoble - Hôpital Sud, Grenoble
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - Groupe Hospitalier du Havre - Hôpital J.Monod, Le Havre
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Centre Hospitalier du Mans, Le Mans
  - Polyclinique de Riaumont, Liévin
  - CHRU Lille - Hôpital Salengro, Lille
  - CHU de Limoges, Limoges
  - CH Saint Philibert, Lomme
  - Hôpital de la Conception, Marseille
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHU Montpellier, Hôpital Lapeyronie, Montpellier
  - Centre Hospitalier de Mulhouse - Hôpital Emile Muller, Mulhouse
  - CHU de Nantes - Hôtel Dieu, Nantes
  - CHU de Nice - Hôpital de l'Archet 1, Nice
  - Centre Hospitalier Régional d'Orléans, Hôpital de la Source, Orléans
  - CHU Chenevier - Mondor, Paris
  - Groupe Hospitalier Diaconesses - Hôpital de la Croix Saint-Simon, Paris
  - Hôpital Bichat, Paris
  - Hôpital de la Pitié Salpétrière, Paris
  - Hôpital Lariboisière, Paris
  - Hôpital Saint-Antoine, Paris
  - CHU de Poitiers - Hôpital de la Milétrie, Poitiers
  - Centre Hospitalier René Dubos, Pontoise
  - CHU de Reims - Hôpital Maison Blanche, Reims
  - CHU de Rennes - Hôpital Sud, Rennes
  - CHU de Rouen - Hôpital Bois Guillaume, Rouen
  - CHU de Saint-Etienne, Saint-Etienne
  - Hôpital de Hautepierre, Strasbourg
  - CHU de Toulouse - Hôpital Purpan, Toulouse
  - CHU de Nancy - Hôpital Brabois, Vandœuvre-lès-Nancy
- Centre Hospitalier - Princesse Grâce de Monaco, Monaco, Monaco

REFERENCES:
- [Result] Gottenberg JE, Brocq O, Perdriger A, Lassoued S, Berthelot JM, Wendling D, Euller-Ziegler L, Soubrier M, Richez C, Fautrel B, Constantin AL, Mariette X, Morel J, Gilson M, Cormier G, Salmon JH, Rist S, Liote F, Marotte H, Bonnet C, Marcelli C, Sellam J, Meyer O, Solau-Gervais E, Guis S, Ziza JM, Zarnitsky C, Chary-Valckenaere I, Vittecoq O, Saraux A, Pers YM, Gayraud M, Bolla G, Claudepierre P, Ardizzone M, Dernis E, Breban MA, Fain O, Balblanc JC, Aberkane O, Vazel M, Back C, Candon S, Chatenoud L, Perrodeau E, Sibilia J, Ravaud P. Non-TNF-Targeted Biologic vs a Second Anti-TNF Drug to Treat Rheumatoid Arthritis in Patients With Insufficient Response to a First Anti-TNF Drug: A Randomized Clinical Trial. JAMA. 2016 Sep 20;316(11):1172-1180. doi: 10.1001/jama.2016.13512. PMID 27654603
- [Derived] Nguyen MVC, Courtier A, Adrait A, Defendi F, Coute Y, Baillet A, Guigue L, Gottenberg JE, Dumestre-Perard C, Brun V, Gaudin P. Fetuin-A and thyroxin binding globulin predict rituximab response in rheumatoid arthritis patients with insufficient response to anti-TNFalpha. Clin Rheumatol. 2020 Sep;39(9):2553-2562. doi: 10.1007/s10067-020-05030-6. Epub 2020 Mar 24. PMID 32212002
- [Derived] Virone A, Bastard JP, Fellahi S, Capeau J, Rouanet S, Sibilia J, Ravaud P, Berenbaum F, Gottenberg JE, Sellam J. Comparative effect of tumour necrosis factor inhibitors versus other biological agents on cardiovascular risk-associated biomarkers in patients with rheumatoid arthritis. RMD Open. 2019 Jul 21;5(2):e000897. doi: 10.1136/rmdopen-2019-000897. eCollection 2019. PMID 31413865
- [Derived] Riviere E, Sellam J, Pascaud J, Ravaud P, Gottenberg JE, Mariette X. Serum IL-33 level is associated with auto-antibodies but not with clinical response to biologic agents in rheumatoid arthritis. Arthritis Res Ther. 2018 Jun 8;20(1):122. doi: 10.1186/s13075-018-1628-6. PMID 29884223